CLINICAL TRIAL: NCT01935401
Title: Self-regulatory Control and Eating: A Neuroimaging Study of Bulimia Nervosa
Status: Completed | Type: Observational
Sponsor: Michael Lowe (Other)
Responsible Party: Sponsor-Investigator, Michael Lowe, PI, Drexel University
Organization: Drexel University (Other)
Other Study IDs: 1F31MH097406 (NIH)
Record Dates: First submitted 2013-08-05; First posted 2013-09-05 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Bulimia Nervosa
Keywords: Bulimia Nervosa; Bulimia; Response Inhibition; fNIR; Neuroimaging
MeSH Terms: conditions — Bulimia Nervosa; Bulimia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Women with Bulimia Nervosa: fNIR
  - Functional near-infrared spectroscopy measured-brain activity
- Healthy Controls: fNIR
  - Functional near-infrared spectroscopy measured-brain activity

SUMMARY:
The purpose of this study will be to replicate previous findings of deficits in prefrontal activation during response inhibition tasks in bulimia nervosa and extend these findings by demonstrating similar deficiencies in activity during a functional behavioral task that requires the inhibition of eating. Findings from this study will potentially help to elucidate the underlying neural mechanisms of bulimia nervosa, and thus inform treatment and prevention efforts.

DETAILED DESCRIPTION:
Bulimia nervosa (BN), is a serious psychiatric disorder that has high rates of comorbidity and often results in role impairment for the suffer. Thus far, although psychosocial and behavioral risk factors and correlates of BN have been extensively researched, relatively few studies have focused on brain-based determinants of BN. Identification of neural mechanisms associated with self-regulatory control that may be integral in the development, maintenance, and prevention of this debilitating condition would better inform treatment development and eating disorder prevention efforts.

Participation in this study consists of a 3-3.5 hours study visit as well a a one year follow up visit. The first portion of initial study visit is part of the screening process, in which individuals will complete several questionnaires and be interviewed by the study researcher in order to confirm eligibility. If a participant is eligible after the screening portion, they move onto the rest of the initial visit. During the initial visit, participants will complete a button pressing go/no-go task as well as a sipping go/no-go task, all while wearing a functional near-infrared spectroscopy (fNIR) device.

At a one year follow up appointment, individuals will again complete a variety of self-report questionnaires and be interviewed by the study researcher, thus completing the same measures used as screening tools in the initial visit.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Right-handed
* Age 18-45
* Between 85 and 120% of ideal body weight based on height
* Currently meeting proposed DSM-5 criteria for Bulimia Nervosa (at least one objective bulimic episode and compensatory purging episode per week for the past three months)
* Purging via self-induced vomiting
* Duration of illness of at least 6 months

Exclusion Criteria:

* Current significant medical illness
* Any disorder or condition resulting in difficulty swallowing (e.g., dysphagia)
* History of neurological disorders or diseases (e.g., stroke, seizures, heart disease, head trauma with loss of consciousness)
* Drug or alcohol abuse in the past 6 months or any history of alcohol or drug dependence
* Use of marijuana or any other illegal drug (e.g., cocaine, heroin, ecstasy) in the week before the study visit
* IQ less than 75
* Pregnancy, lactation, or planning to become pregnant in the next year
* Allergy to sucrose, dairy, wheat, gluten, apples (i.e., any of the ingredients in the strawberry yogurt shake or in the standardized meal prior to study participation)
* Participants rating the strawberry yogurt shake as a 5 or lower on a 9-point category scale of liking will be excluded from further study
* Meeting the criteria for a diagnosis of Attention Deficit Hyperactivity Disorder
* Any other current major Axis I disorder, other than major depressive disorder (MDD) or generalized anxiety disorder (GAD)
* Inability to consent
* Prisoner

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women (ages 18-45 years) with bulimia nervosa and age, BMI, and IQ-matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2011-06; Primary Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Functional near-infrared spectroscopy | Day 1

SECONDARY OUTCOMES:
Body mass index | Day 1 and 1 year
  Body mass index, calculated from height and weight measurements
Eating disorder examination (EDE) | Day 1 and 1 Year
  Used to assess eating disorder symptom frequency and severity, including binge eating episode frequency.
Wechsler Abbreviated Scale of Intelligence (WASI™) | Day 1
Mini-International Neuropsychiatric Interview (MINI) | Day 1
Button pressing go/no-go task | Day 1
Go/no-go sipping task | Day 1
Psychosocial self-report measures | Day 1 and 1 Year
  Measures to be administered include: Power of Food Scale (PFS), Beck Anxiety Inventory (BAI), Center for Epidemiological Studies Depression Scale (CES-D), Barratt Impulsivity Scale, Version 11 (BIS), Eating Loss of Control Scale (ELOCS), Difficulties in Emotion Regulation Scale (DERS), and Behavioral Inhibition and Behavioral Activation (BIS/BAS) Scales
Positive and Negative Affect Schedule (PANAS) | Day 1
  This measure will assess mood ratings before the participant completes the standard go/no-go task and the sipping go/no-go task
Generalized Labeled Magnitude Scale (gLMS) | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Lowe, Ph.D., Principal Investigator — Drexel University
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States